CLINICAL TRIAL: NCT02063126
Title: A Randomized, Double-blind, Placebo-controlled, Comparative Clinical Trial to Measure the Maximun Heart Rate During a Cycle Ergometer Test After ReConnect® Supplementation in CFS.
Brief Title: Clinical Trial to Measure the Maximun HR After ReConnect ® Supplementation vs. Placebo in CFS.
Acronym: ReConnect
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: VITAE NATURAL NUTRITION, S.L. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VITAE 01-2012
Record Dates: First submitted 2014-02-05; First posted 2014-02-14 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Coenzyme Q10 plus NADH; maximum Heart Rate; Fatigue; Pain; Sleep
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Pain | interventions — NAD; coenzyme Q10; Phosphoserine; Serine; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReConnect (Active Comparator): CFS patients who were randomized to measure the effect of oral ReConnect supplementation (NADH: 20 mg/day, Coenzyme Q10: 200 mg/day; 4 tablets/day) on the maximum HR during 8-weeks in term.
  Interventions: Dietary Supplement: ReConnect (NADH plus CoQ10)
- Placebo (Placebo Comparator): CFS patients who were randomized to measure the effect of oral Placebo supplementation ( phosphoserine and vitamin C, 4 tablets/day) on the maximum HR during 8-weeks in term.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ReConnect (NADH plus CoQ10) — ReConnect supplementation (NADH: 20 mg/day plus CoQ10: 200mg/day) divided into two daily dose ( 2 tablets/ before breakfast and 2 tablets/ before lunch)
  Placebo supplementation divided into two daily dose ( 2 tablets/ before breakfast and 2 tablets/ before lunch)
  Other Names: Placebo
  Arms: ReConnect
Dietary Supplement: placebo — placebo (phosphoserine/serine plus vitamin C) supplementation divided in two daily doses (2 tablets/before brekfast and 2 tablets/before lunch)
  Other Names: Placebo (phosphoserine/serine plus vitamin C)
  Arms: Placebo

SUMMARY:
The main objective is evaluate to safety and efficacy of oral Reconnect ® (food supplementation composed by Coenzyme Q10, NADH, phosphoserine y vitamin C) on the maximum HR during an exercise test in CFS

DETAILED DESCRIPTION:
Chronic Fatigue Syndrome (CFS) is a serious, complex and extremely debilitating chronic illness, but often misunderstood characterized by prolonged fatigue, the hallmark of the condition and multiple nonspecific symptoms. The World Health Organization has recognized CFS as a disease that affecting the nervous system (ICD-10 G93.3) and multiple body systems. The etiology is unknown. Previous studies have demonstrated in CFS patients a significant reduction in plasma and intracellular Peripheral Blood Mononuclear Cells concentrations of Coenzyme Q10 and NADH, which correlate with clinical symptoms of the disease. Hypothesis: Supplementation with CoQ10 plus NADH could be beneficial in the improvement of clinical and molecular parameters in this disease. The primary endpoint is to evaluate the efficacy of oral Reconnect ® suplementation on the maximum heart rate changes during an exercise test in CFS. The secondary endpoints are to evaluate the effect of Reconnect ® suplementation on perception of fatigue (assessed by FIS), pain (McGill Pain Index Questionnaire), and sleep disruption (Pittsburgh Sleep Index Questionnaire).

Patients and Methods: A total of 80 consecutive women patients with a diagnosis of CFS according to the 1994 CDC Fukuda's definition criteria were initially evaluated and enrolled in this study. The majority were excluded for no meet the inclusion criteria of the study. All subjects are treatment with ReConnect® containing CoQ10 plus NADH versus placebo. Fatigue levels, pain and sleep disturbances are scored using the Fatigue Impact Scale, McGill Pain Questionnaire and Pittsburgh Sleep Quality Index, respectively.

Discussion: To our knowledge, no previous studies have yet evaluated the effectiveness of oral ReConnect supplementation in CFS. ReConnect containing the combination of CoQ10 plus NADH and other nutrients (phosphoserine and Vitamin C) can help to improve clinical symptoms and restore mitochondrial function and oxidative stress reducing fatigue, pain and sleep impairments in CFS. The combination of these supplements can result in a safe and effective therapy to reduce fatigue, pain and improve sleep as well help restore quality of life of CFS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients female between 18 and 65 years old.
* CFS patients diagnosed with Chronic Fatigue Syndrome (CFS Clinical Unit, Vall d'Hebron Hospital, Barcelona, Spain)
* Heart rate in radial pulse and seated between 50 to100 bpm, systolic BP between 100 to 140 mm Hg and diastolic BP between 50 to 90 mm Hg.
* Patients who give a written informed consent before initiating the study.

Exclusion Criteria:

* Patients for that is contraindicated or is not advisable to carry-out an ergometer exercise test.
* Patients who are participating in another clinical trial of the same or differents nature in the last 30 days prior to inclusion.
* Any participants who, in the opinion of the investigator, may not be able to follow instructions or make a good treatment compliance.
* Subjects that do not give written informed consent to participate in the study.
* Participants who are receiving any drug or banned substances and is expected that withdrawal of some medications/products not allowed in the study involves a significants problem.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum HR changes after ReConnect supplementation during an incremental exercise test in CFS patients | within the first 30 days (plus or minus 15 days) after treatment
  Researchers hypothesize that the low maximun HR in CFS is tied to the brain via the autonomic nervous system, which regulates the body's automatic functions. Dysregulation of the autonomic nervous system is called dysautonomia and is believed to be a feature of CFS patients.

SECONDARY OUTCOMES:
Perception of fatigue, pain and sleep disruption after ReConnect supplementation during an incremental exercise test in CFS patients | within the first 30 days (plus or minus 15 days)
  Researchers hypothesize that perception of fatigue, pain and sleep disturbances in CFS is tied to the brain via the autonomic nervous system, which regulates the body's automatic functions. Dysregulation of the autonomic nervous system is called dysautonomia and is believed to be a feature of CFS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alegre-Martin, MD, PhD, Principal Investigator — Vall d'Hebron University Hospital Research Institute. Internal Medicine Unit.
Locations (1):
- Vall Hebron University Hospital, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Castro-Marrero J, Saez-Francas N, Segundo MJ, Calvo N, Faro M, Aliste L, Fernandez de Sevilla T, Alegre J. Effect of coenzyme Q10 plus nicotinamide adenine dinucleotide supplementation on maximum heart rate after exercise testing in chronic fatigue syndrome - A randomized, controlled, double-blind trial. Clin Nutr. 2016 Aug;35(4):826-34. doi: 10.1016/j.clnu.2015.07.010. Epub 2015 Jul 17. PMID 26212172
- [Derived] Castro-Marrero J, Cordero MD, Segundo MJ, Saez-Francas N, Calvo N, Roman-Malo L, Aliste L, Fernandez de Sevilla T, Alegre J. Does oral coenzyme Q10 plus NADH supplementation improve fatigue and biochemical parameters in chronic fatigue syndrome? Antioxid Redox Signal. 2015 Mar 10;22(8):679-85. doi: 10.1089/ars.2014.6181. Epub 2014 Dec 18. PMID 25386668